CLINICAL TRIAL: NCT00749970
Title: Validity of the Spanish Version of Subjective Well-being Under Neuroleptics Scale (SWN-K) in Patients With Schizophrenia
Acronym: SWN-K
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Diez, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2008/1
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: schizophrenia; subjective well-being; psychometric validation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Observational, short-term prospective, multicenter study to assess psychometric properties of the Spanish version of SWN-K scale in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder (DSM-IV TR criteria)
* Stabilized out-patients
* Under treatment with an oral antipsychotic drug

Exclusion Criteria:

* Administration of a depot antipsychotic drug
* Participation in another clinical trial within 4 weeks prior to enrolment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient aged 18-year old or older with a diagnosis of schizophrenia, schizoaffective disorder, or shizophreniform disorder
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
SWN-K | 7 days
PANSS | 7 days

SECONDARY OUTCOMES:
CGI-I | 7 days

CONTACTS AND LOCATIONS:
Locations (14):
- Spain (14):
  - Research Site, Alicante
  - Research site, Barcelona
  - Research site, Burgos
  - Research Site, Córdoba
  - Research Site, Granada
  - Research site, Madrid
  - Research Site, Mallorca
  - Research Site, Salamanca
  - Research Site, Seville
  - Research site, Tarragona
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Vitoria-Gasteiz
  - Research Site, Zaragoza